CLINICAL TRIAL: NCT01266005
Title: A Study to Compare and Evaluate Intrahepatic cccDNA Reduction After Administrating Clevudine or Entecavir in the Chronic HBV Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Bukwang, Bukwang Pharm.Co.,LTD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLV-410
Record Dates: First submitted 2010-12-19; First posted 2010-12-24 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis B
Keywords: HBe Ag(-) Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine; entecavir

ARMS (2):
- 1 (Experimental): Clevudine 30mg
  Interventions: Drug: Clevudine
- 2 (Active Comparator): Entecavir 0.5mg
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Clevudine — 30mg,QD
  Other Names: Levovir
  Arms: 1
Drug: Entecavir — 0.5mg QD
  Other Names: Baraclude
  Arms: 2

SUMMARY:
This is a open, randomized, parallel study. Subjects will have Clevudine or Entecavir therapy for 48 weeks(Clevudine:Entecavir = 2:1), and subjects who have Complete Response(HBV DNA negative and ALT normal) will have follow-up period for additional 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is older than 18.
2. Patient who is HBsAg positive for the previous 6 months and with HBV DNA ≥ 1 x 10^5 copies/mL
3. Patient who is HBeAg negative.
4. Patient with ALT≥1×ULN.
5. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Patient is currently receiving antiviral, immunomodulatory, cytotoxic or corticosteroid therapy.
2. Patient is treated with interferon for the previous 6 months.
3. Patient has been treated previously with clevudine, lamivudine, adefovir, entecavir, telbivudine or any other investigational nucleoside for HBV infection.
4. Patient is coinfected with HCV, HDV or HIV.
5. Patient has evidence of ascites, variceal hemorrhage and/or hepatic encephalopathy.
6. Patient has evidence of decompensated Liver cirrhosis and/or hepatocellular carcinoma.
7. Patient has a history of organ transplantation.
8. Patient has the treatment of nephrotoxicity drugs, competitive drugs for kidney to excrete, and/or hepatotoxicity drugs for the previous 2 months from screening.
9. Patient is pregnant or breast-feeding.
10. Patient has a clinically relevant history of abuse of alcohol or drugs.
11. Patient has a significant immunocompromised, gastrointestinal, renal, hematological, psychiatric, bronchopulmonary, biliary diseases excluding asymptomatic GB stone, neurological, cardiac, oncologic, allergic disease or medical illness that in the investigator's opinion might interfere with therapy. The patient with a benign tumor, excluded if judged by an investigator that the continuation of study would be interfered by the tumor.
12. Patient has creatinine clearance less than 60mL/min as estimated by the following formula: (140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Intrahepatic cccDNA reduction from baseline | week 48

SECONDARY OUTCOMES:
Proportion of patients with HBV DNA below LOD by real-time PCR | day1(predose), every 12 weeks during treatment period(48weeks), every 8 weeks during follow-up period(48weeks)
Reduction of HBV DNA level from baseline | day1(predose), every 12 weeks during treatment period(48weeks), every 8 weeks during follow-up period(48weeks)
ALT normalization | day1(predose), every 12 weeks during treatment period(48weeks), every 8 weeks during follow-up period(48weeks)
Reduction of sAg titer from baseline | day1(predose), every 12 weeks during treatment period(48weeks), every 8 weeks during follow-up period(48weeks)
Proportion of maintaining sustained effect | every 8 weeks during follow-up period(48weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- 9 Sites, Seoul, South Korea